CLINICAL TRIAL: NCT04804592
Title: Investigation in Variability and Repeatability of Corneal Sensation in a Normal Population and Contact Lens Wearers
Brief Title: Investigation in Corneal Sensation and Contact Lens Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Nosch (Other)
Responsible Party: Sponsor-Investigator, Daniela Nosch, Professor, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-00438
Record Dates: First submitted 2021-03-11; First posted 2021-03-18 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Cornea; Sense Loss; Cornea
Keywords: cornea; ocular surface sensation; corneal sensitivity; contact lens wear
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: SiHy CL (Experimental): Silicone hydrogel (SiHy) CL wear at least 3 days per week and at least 8 hours per day;
  Interventions: Device: Tactile Esthesiometer Prototype; Device: Liquid Jet Esthesiometer Prototype; Device: Cochet Bonnet esthesiometer
- Group B: RGP CL (Experimental): Rigid gas permeable (RGP) CL wear at least 3 days per week and at least 8 hours per day;
  Interventions: Device: Tactile Esthesiometer Prototype; Device: Liquid Jet Esthesiometer Prototype; Device: Cochet Bonnet esthesiometer
- Group C: no CL wear (Experimental): No current CL wear for at least 3 months;
  Interventions: Device: Tactile Esthesiometer Prototype; Device: Liquid Jet Esthesiometer Prototype; Device: Cochet Bonnet esthesiometer

INTERVENTIONS:
Device: Tactile Esthesiometer Prototype — A round plastic nozzle (1.8mm diameter) used as a stimulus for corneal sensation threshold measurement
Device: Liquid Jet Esthesiometer Prototype — Balanced salt solution with a pH value similar to the tear film uesd as a liquid jet stimulus for corneal sensation threshold measurement
Device: Cochet Bonnet esthesiometer — A nylon thread (0.12mm diameter) used as a stimulus for corneal sensation threshold measurement

SUMMARY:
The aim is to find out more about how corneal sensory fibres react to different types of stimuli (liquid / tactile / nylon thread) and how this can be consciously perceived by the individual. Is it possible to generate a stimulus that delivers a repeatable and reliable response within a useful stimulus force range which allows an interpretation / evaluation of normal / expected activity of superficial nerve fibres in the cornea? The study group will be divided into three groups of individuals: two groups with different types of contact lenses (CL) and one without CL, as sensitivity changes are thought to occur with CL wear. A very interesting research question is to find out, if such sensitivity differences can be detected with the nature of the stimuli applied in this study.

DETAILED DESCRIPTION:
The aim of this study is to gain more physiological knowledge about ocular surface sensation (corneal sensitivity), with application of three different concepts employing different types of stimuli for triggering a response from the pain sensitive nerve endings in the superficial cornea: 1) tactile method: a round plastic nozzle (2 mm diameter) is applied to the ocular surface with a defined, low force for a duration of 100ms. 2) liquid jet method: a liquid jet (isotonic saline) of a temperature to match ocular surface temperature is applied to the ocular surface with low pressure and low volume, from a distance of 15 mm.3) commercially available Cochet Bonnet esthesiometer (nylon thread). The study group will be divided into three groups of individuals: two groups with different types of contact lenses (CL) and one without CL, as sensitivity changes are thought to occur with CL wear. A very interesting research question is to find out, if such sensitivity differences can be detected with the nature of the stimuli applied in this study.

Current knowledge about human corneal sensitivity is limited, as applied methods for ocular surface sensation measurement are limited with regards to reproducibility / accuracy.

Corneal sensitivity represents a neurological response from the free nerve endings within the epithelium. They are sensitive to mechanical, electrical, chemical or thermal stimuli and hence have a protective function for the cornea. Corneal nerves play an important role in cell growth and proliferation of epithelial cells, wound healing and repair. In experimental studies, corneal denervation has been reported to result in epithelial changes: increased permeability, decreased proliferation, changed appearance and delayed wound healing. Therefore, intact corneal innervation is required to maintain the integrity of a normal corneal epithelium. Corneal sensory nerves are believed to play an important role in maintaining the resting tear flow, as their afferent impulses from the ocular surface lead to a reflex response, best described by the lacrimal functional unit: an integrated system comprising the ocular surface tissues (cornea, corneal limbus, conjunctiva, conjunctival blood vessels, and eyelids), the tear secreting components (main and accessory lacrimal glands, meibomian glands, conjunctival goblet, and epithelial cells), and the sensory and motor nerves that connect them.

Current knowledge about ocular surface sensitivity is insufficient, as currently available measurement possibilities lack repeatability and accuracy. Before a new instrument can be developed, more research is required, in order to find a suitable concept for precise sensitivity measurement. For this purpose, two new different concepts with different / new stimulus types will be applied repeatably on healthy eyes in this study. The aim is to find out more about how corneal sensory fibres react to different types of stimuli (liquid / tactile / nylon thread) and how this can be consciously perceived by the individual. Is it possible to generate a stimulus that delivers a repeatable and reliable response within a useful stimulus force range which allows an interpretation / evaluation of normal / expected activity of superficial nerve fibres in the cornea? The study group will be divided into three groups of individuals: two groups with different types of contact lenses (CL) and one without CL, as sensitivity changes are thought to occur with CL wear.

ELIGIBILITY:
Inclusion Criteria:

Group A:

Silicone hydrogel (SiHy) CL wear at least 3 days per week and at least 8 hours per day; 18 - 50 years of age; healthy eyes with OSDI </= 13

Group B:

Rigid gas permeable (RGP) CL wear at least 3 days per week and at least 8 hours per day; 18 - 50 years of age; healthy eyes with OSDI </= 13

Group C:

No current CL wear for at least 3 months; 18 - 50 years of age; healthy eyes with OSDI </= 13

Exclusion Criteria:

* Systemic disease that may affect ocular health, such as diabetes
* Injury and history of operations on the anterior segment of the eye
* regular application of systemic or ocular medication known to affect the tear film, specifically on the day of measurement

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Repeatability of mechanical corneal sensation thresholds with the liquid jet protoype esthesiometer | two weeks
  Evaluation of repeatability of mechanical corneal sensation thresholds for the measurement with the liquid jet esthesiometer prototype instrument (in mbar): the corneal sensation thresholds will be obtained with the double staircase method (with forced choice) and the stimulus represents a liquid jet (consisting of isotonic saline solution).
Repeatability of mechanical corneal sensation thresholds with the tactile prototype esthesiometer | two weeks
  Evaluation of variability / repeatability of mechanical corneal sensation thresholds for the measurement with the tactile esthesiometer prototype instrument (in mN): the corneal sensation thresholds will be obtained with the double staircase method (with forced choice) and the stimulus represents a small, round plastic ball.
Repeatability of mechanical corneal sensation thresholds with the Cochet Bonnet esthesiometer | two weeks
  Evaluation of repeatability of mechanical corneal sensation thresholds for the measurement with the Cochet Bonnet instrument (in mN): the corneal sensation thresholds will be obtained with the double staircase method (with forced choice) and the stimulus represents a nylon thread, whereby its force is proportional to the length of the nylon thread applied to the corneal surface.

SECONDARY OUTCOMES:
Correlation between corneal sensation thresholds with the Cochet Bonnet esthesiometer | one day
  Correlation between corneal sensitivity thresholds (in mN) obtained with the Cochet Bonnet esthesiometer
Correlation between corneal sensation thresholds with the liquid jet prototype esthesiometer | one day
  Correlation between corneal sensitivity thresholds (in mbar) obtained with the liquid jet prototype esthesiometer
Correlation between corneal sensation thresholds with the tactile prototype esthesiometer | one day
  Correlation between corneal sensitivity thresholds (in mN) obtained with the tactile prototype esthesiometer
Comparison of corneal sensation thresholds, obtained with the Cochet Bonnet esthesiometer, between the three groups in the study population | two weeks
  Comparison of corneal sensation thresholds obtained with the Cochet Bonnet esthesiometer between the three groups in the study population
Comparison of corneal sensation thresholds, obtained with the liquid jet prototype esthesiometer, between the three groups in the study population | two weeks
  Comparison of corneal sensation thresholds, obtained with the liquid jet prototype esthesiometer, between the three groups in the study population
Comparison of corneal sensation thresholds, obtained with the tactile prototype esthesiometer, between the three groups in the study population | two weeks
  Comparison of corneal sensation thresholds, obtained with the tactile prototype esthesiometer, between the three groups in the study population

CONTACTS AND LOCATIONS:
Overall Officials: Daniela S Nosch, PhD, Principal Investigator — University of Applied Sciences and Arts Northwestern Switzerland FHNW
Locations (1):
- Institute of Optometry, FHNW, Olten, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belmonte C, Acosta MC, Gallar J. Neural basis of sensation in intact and injured corneas. Exp Eye Res. 2004 Mar;78(3):513-25. doi: 10.1016/j.exer.2003.09.023. PMID 15106930
- [Background] Bergenske PD, Polse KA. The effect of rigid gas permeable lenses on corneal sensitivity. J Am Optom Assoc. 1987 Mar;58(3):212-5. PMID 3471806
- [Background] Knoll HA, Williams J. Effects of hydrophilic contact lenses on corneal sensitivity. Am J Optom Arch Am Acad Optom. 1970 Jul;47(7):561-3. doi: 10.1097/00006324-197007000-00007. No abstract available. PMID 5270397
- [Background] Millodot M. Does the long term wear of contact lenses produce a loss of corneal sensitivity? Experientia. 1977 Nov 15;33(11):1475-6. doi: 10.1007/BF01918817. PMID 923715
- [Background] Muller LJ, Marfurt CF, Kruse F, Tervo TM. Corneal nerves: structure, contents and function. Exp Eye Res. 2003 May;76(5):521-42. doi: 10.1016/s0014-4835(03)00050-2. PMID 12697417
- [Background] Golebiowski B, Chao C, Stapleton F, Jalbert I. Corneal Nerve Morphology, Sensitivity, and Tear Neuropeptides in Contact Lens Wear. Optom Vis Sci. 2017 Apr;94(4):534-542. doi: 10.1097/OPX.0000000000001063. PMID 28338565
- [Background] Stapleton F, Chao C, Golebiowski B. Topical Review: Effects of Contact Lens Wear on Corneal, Conjunctival, and Lid Margin Sensitivity. Optom Vis Sci. 2019 Oct;96(10):790-801. doi: 10.1097/OPX.0000000000001429. PMID 31592962
- [Background] Golebiowski B, Papas EB, Stapleton F. Factors affecting corneal and conjunctival sensitivity measurement. Optom Vis Sci. 2008 Apr;85(4):241-6. doi: 10.1097/OPX.0b013e3181694f96. PMID 18382334
- [Background] Stapleton F, Golebiowski B, Skotnitsky C, Tan ME, Holden BA. Corneal and conjunctival sensitivity in intolerant contact lens wearers. J Optom. 2015 Jan-Mar;8(1):62-3. doi: 10.1016/j.optom.2014.05.004. Epub 2014 Jun 7. No abstract available. PMID 25649641
- [Background] Golebiowski B, Papas EB, Stapleton F. Corneal and conjunctival sensory function: the impact on ocular surface sensitivity of change from low to high oxygen transmissibility contact lenses. Invest Ophthalmol Vis Sci. 2012 Mar 9;53(3):1177-81. doi: 10.1167/iovs.11-8416. PMID 22281824